CLINICAL TRIAL: NCT04418557
Title: COVID-19 and Obstetric Transmission
Acronym: COVIDOB
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Cuyahoga County Board of Health (Unknown); The Cleveland Clinic (Other); MetroHealth Medical Center (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Rachel Pope, Assistant Professor, University Hospitals Cleveland Medical Center
Other Study IDs: 20200479
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID; Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Maternal blood, neonatal blood, amniotic fluid, amnion, chorion, umbilical cord, vaginal secretion, cord blood, newborn throat swab, breastmilk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant women without COVID-19 Infection: Women who are tested for COVID-19 at the time of admission for labor and delivery and test negative
  Interventions: Diagnostic Test: RT-PCR and antibody testing
- Pregnant women with a history of COVID-19 infection: Women who are tested for COVID-19 at any point during their pregnancy, including at the time of admission for labor and delivery, and test positive
  Interventions: Diagnostic Test: RT-PCR and antibody testing
- Pregnant women vaccinated for COVID-19: Women who are vaccinated against COVID-19 at any point during their pregnancy

INTERVENTIONS:
Diagnostic Test: RT-PCR and antibody testing — Testing of amniotic fluid, cord blood, amnion and chorion, umbilical cord, vaginal mucous, maternal and neonatal sera, neonatal throat swab, and breast milk.
  Groups: Pregnant women with a history of COVID-19 infection; Pregnant women without COVID-19 Infection

SUMMARY:
The aim of this study is to capture data, laboratory markers, and clinical outcomes of obstetric and neonatal outcomes in cases of COVID-19 during pregnancy and of pregnancies exposed to a COVID-19 vaccine in Cuyahoga County.

DETAILED DESCRIPTION:
A review of the 55 cases of obstetric COVID-19 cases world-wide demonstrate the following fetal complications of COVID-19: miscarriage (2%), intrauterine growth restriction (IUGR; 10%), pre-eclampsia, and pre-term birth (39%). In Wuhan, China, nine women who were COVID-19 positive were surveilled for vertical transmission and overall obstetric and early neonatal outcomes. Amniotic fluid, umbilical cord blood, and neonatal throat swabs were collected at the time of delivery, and breastmilk samples were collected after lactation commenced. There was no viral detection of COVID-19 demonstrated.2 However, two neonates in the United Kingdom have tested positively for COVID-19 after delivery from an infected mother. Most recently, antibodies were detected (IgM and IgG) in the serum of a neonate born via cesarean delivery to a known positive mother. Therefore, vertical transmission has not been completely ruled out.

Additionally, infection at varying times of pregnancy has not been well delineated or correlated to neonatal or maternal outcomes at time of delivery. Therefore, there is a need to continue surveying and documenting clinical findings in obstetric COVID-19 cases.

This study will follow pregnant women who are diagnosed during any point of their pregnancy with COVID-19 and those who were vaccinated. during pregnancy. The aim will be to evaluate maternal and neonatal specimens for the presence of COVID-19 virus, immune and cellular response.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection at any time of the pregnancy, or presumed case by symptoms and direct contact with a positive case
* Pregnancy documented by ultrasound

Exclusion Criteria:

* COVID-19 infection before or after pregnancy
* Person under investigation, but not a presumed or known positive case

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — must be pregnant
Study Population: Pregnant women who have been diagnosed with COVID-19 at any point of their pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Presence of COVID-19 virus | At time of delivery
  Viral presence in any of the collected specimens

SECONDARY OUTCOMES:
Presence of antibodies to COVID-19 virus | At time of delivery and 24 hours of life of the newborn
  Antibodies detected in any of the collected specimens

OTHER OUTCOMES:
Immune responses to COVID-19 virus What is the Immune responses of a mother infected with COVID-19 and neonates? What is the Immune responses of a mother infected with COVID-19 and neonates? Immune response to COVID-19 virus | At time of delivery and 24 hours of life of the newborn
  Innate/Adaptive cell function and immune response

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dong L, Tian J, He S, Zhu C, Wang J, Liu C, Yang J. Possible Vertical Transmission of SARS-CoV-2 From an Infected Mother to Her Newborn. JAMA. 2020 May 12;323(18):1846-1848. doi: 10.1001/jama.2020.4621. PMID 32215581
- [Result] Chen H, Guo J, Wang C, Luo F, Yu X, Zhang W, Li J, Zhao D, Xu D, Gong Q, Liao J, Yang H, Hou W, Zhang Y. Clinical characteristics and intrauterine vertical transmission potential of COVID-19 infection in nine pregnant women: a retrospective review of medical records. Lancet. 2020 Mar 7;395(10226):809-815. doi: 10.1016/S0140-6736(20)30360-3. Epub 2020 Feb 12. PMID 32151335